CLINICAL TRIAL: NCT07376694
Title: Improving Uptake of Bowel Cancer Screening Among South Asian Adults in Bradford
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hull (Other)
Collaborators: Bradford Teaching Hospitals NHS Foundation Trust (Other Government); Gateshead Health NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Lesley Smith, Professor, University of Hull
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: RS213-332905
Record Dates: First submitted 2026-01-12; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-11

CONDITIONS: Bowel Cancer Screening
Keywords: Screening; FOBT; non-randomised trial; South Asian; FIT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced screening kit (Experimental): Culturally tailored enhanced screening kit, comprising an instruction letter and booklet, and a bio-degradable poo catcher
  Interventions: Other: Bowel cancer screening kit
- Usual kit (Active Comparator): Screening kit only
  Interventions: Other: Bowel cancer screening kit

INTERVENTIONS:
Other: Bowel cancer screening kit — Home Fecal Occult Blood Test kit
  Other Names: FOBT

SUMMARY:
Bowel cancer is the second most common cause of cancer related deaths in England. Bowel cancer screening can reduce bowel cancer deaths by detecting bowel cancer early. Previous research has shown that screening can lower a person's risk of dying from bowel cancer by over 25%. In England, the NHS offers free bowel cancer screening for adults aged 60 - 74 years who are registered with a GP every two years, but screening uptake remains poor among those in deprived areas and amongst minority ethnic groups. In socioeconomically deprived areas like Bradford, where there is a high proportion of South Asian residents, bowel cancer screening uptake is low compared to other parts of England. The investigators previous research has shown that people of South Asian ethnicity are limited by many factors beyond language barriers and thus require culturally tailored approaches to facilitate uptake.

For this study, the investigators will aim to answer the question: 'Does a culturally tailored enhanced screening kit, comprising an instruction letter and booklet, and a bio-degradable poo catcher increase bowel cancer screening uptake among South Asians living in Bradford?'. Over a 6-month period, individuals registered in 17 GP practices in Bradford and due to receive their NHS bowel cancer screening invitation will be assigned to two groups: standard kit (usual screening kit only) and enhanced kit (culturally tailored instruction letter and biodegradable poo catcher). Uptake of bowel cancer screening among South Asian participants in each group will be assessed 13 weeks after the identification of the final participant. The findings of this study will provide valuable information for policy makers about how to address population specific barriers to bowel cancer screening using culturally tailored approaches in the UK.

DETAILED DESCRIPTION:
Bowel cancer is the fourth most common cancer and the second leading cause of cancer deaths in England [1,2]. Screening can improve survival by detecting cancer earlier, when cancer is easier to treat [3]. However, participation in screening is sub-optimal, and there are ethnic and regional inequalities in uptake [4]. Indeed, in 2022, uptake of bowel cancer screening in Yorkshire and Humber was 72.2% overall, but only 67.8% in Bradford [5], where there is a high proportion of South Asian residents (uptake of bowel cancer screening in England has been shown to be 50% lower among South adults, compared with White British adults) [6].

Universal approaches attempting to increase the uptake of bowel cancer screening, such as text-message reminders, have been shown to be effective, but tend to be inaccessible to those whose first language is not English and, thus, may widen health inequalities [7]. In addition, recent research indicates that a plethora of culturally specific barriers, over and above language barriers, prohibit participation in bowel cancer screening by South Asian individuals [8,9]. Thus, culturally tailored approaches, which address population-specific barriers, are needed to ensure equitable access to, and uptake of, screening.

The investigators have spent the past two years working with South Asian communities to understand their barriers to participation, and have identified the following barriers to completing the test: 1) lack of knowledge about bowel cancer and screening (knowledge); 2) lack of language, literacy and physical ability (skills) to carry out the home test; 3) confidence to carry it out correctly (belief about capabilities); 4) appropriate space and time to carry out the test (environmental context and resources); 5) putting off undertaking the test (memory attention and decision processes); 6) risk perception and fear of cancer (emotions) [8,9].

Mapping previous findings onto the Theoretical Domains Framework (in red) [10] and, subsequently, the Behaviour Change Technique Taxonomy (BCTT) [11], research suggests that interventions which include 'education/information', 'persuasion', 'modelling' and 'enablement' functions (as defined by the BCTT) could address the barriers and increase the completion rate of the home-based bowel cancer screening test (among South Asian adults).

To address the identified barriers, and implement the above functions (in blue) the investigators propose a multifaceted intervention, comprising: 1) an easy to use and hygienic biodegradable poo catcher compared with the standard faecal immunochemical test kit (enablement) [see Appendix A]; 2) an instruction letter and booklet, with additional information on bowel cancer and screening, provided in English and multiple South Asian languages (enablement and education/information); 3) links to YouTube videos on how to use the biodegradable poo catcher (modelling and persuasion) [see Appendix A].

ELIGIBILITY:
Inclusion Criteria:

1. Patients registered with one of 17 participating GP practices in Bradford
2. Patients invited for bowel cancer screening during the implementation period

Exclusion Criteria:

1) Individuals who are self-referrals 2) Type 2 objectors

-

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2300 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Return of bowel screening kit for testing | 13 weeks (screening episode)
  % of individuals who return their bowel screening kit for foecal immunochemical testing measured using data recorded in their clinical records

SECONDARY OUTCOMES:
Bowel cancer screening test result | 13 weeks (screening episode)
  % of individuals who screen positive for the bowel cancer screening test measured using Foecal Immunochemical Test (FIT) result recorded n clinical records

OTHER OUTCOMES:
Practicality of implementation of the enhanced kit | 13 weeks (screening episode)
  Practicality of implementation of the enhanced kit by screening hub staff measured using qualitative interviews
Costs | 13 weeks (screening episode)
  Costs of implementation of the enhanced kit and its distribution measured using qualitative interviews
Acceptability of implementation of enhanced kit | 13 weeks (screening episode)
  Acceptability to bowelc cancer screening hub staff of implementation of the enhanced kit measured using qualitative interviews

CONTACTS AND LOCATIONS:
Locations (1):
- Northeast Bowel cancer Screening Hub, Gateshead, Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Consent for sharing data has not been sought